CLINICAL TRIAL: NCT06878508
Title: Clincial Use of Implantable Ventricular Assist System for Advanced Heart Failure
Brief Title: DuoCor Ventricular Assist System Early Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_DuoCor
Record Dates: First submitted 2025-03-06; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DuoCor Ventricular Assist System (Experimental)
  Interventions: Device: DuoCor Ventricular Assist System

INTERVENTIONS:
Device: DuoCor Ventricular Assist System — The DuoCor VAS is used to provide hemodynamic support by shareing some or all the workload of the left and right ventricles during the support period.

SUMMARY:
Feasibility study of the DuoCor Ventricular Assist System as a treatment for advanced total heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

1. Requiring a biventricular mechanical circulatory support, defined by either of the following criteria:

   * Persistent total heart failure despite under optimal medical management based on current heart failure practice guidelines. OR
   * Development of refractory right heart failure following left ventricular assist device (LVAD) implantation, unresponsive to pharmacological interventions for right heart failure.
2. Patient has signed the informed consent, has full understanding of procedures, and is committed to following study requirements.

Exclusion Criteria:

1. Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy the investigator will require based upon the patient's health status.
2. Technical obstacles which pose the implantation as unsuitable, obtaining the body type, body surface area, and anatomical conditions related to the planned implantation site, in the judgment of the experienced investigators.
3. Pregnancy.
4. Age > 75 years.
5. Presence of an active, uncontrolled infection.
6. Brain death.
7. History of confirmed, untreated abdominal aortic aneurysm (AAA) or thoracic aortic aneurysm (TAA) > 5 cm in diameter.
8. Irreversible cognitive dysfunction, psychosocial issues, or psychiatric disease, likely to impair compliance with the study protocol and DuoCor VAS management which, in the opinion of the investigator, could interfere with the ability to manage the therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite of survival at 3 months post-implantation | 3 months
  Composite of survival to transplant, recovery (defined as complete/ partial removal or explantation of the DuoCor VAS due to cardiac recovery), or survival with the device at 3 months post-implantation

SECONDARY OUTCOMES:
Hospital redmission rate | 3 months
  Rate of unplanned readmissions to the hospital.
Adverse Events. | 3 months
  Adverse Event as defined in INTERMACS Adverse Events (Definition Date: 10/11/2021)

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
At this moment the IPD is not yet available for access and will be updated when it is ready.